CLINICAL TRIAL: NCT05894213
Title: Prevalence and Factors Associated With Sarcopenia in Pre-retirement Aged Adults With Chronic Non-specific Lower Back Pain
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Songsuda Roongsaiwatana, Principal investigator, Mahidol University
Other Study IDs: COA.MURA2019/733
Record Dates: First submitted 2023-04-07; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Sarcopenia; Chronic Lower Back Pain
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the prevalence of sarcopenia in a pre-retirement group with chronic lower back pain and factors associated between sarcopenia and chronic lower back pain in the pre-retirement group.

ELIGIBILITY:
Inclusion Criteria:

1. Be a person between the ages of 50 - 59 years with or without chronic lower back pain longer than 3 months, but without any dangerous signs of lower back pain, sciatica pain, and neurological disorder.
2. Be able to walk continuously for at least 10 minutes.
3. Give written consent to join the research project.

Exclusion Criteria:

1. Have a history of spinal fracture, spondylolisthesis, scoliosis, or osteomyelitis.
2. Have a neurological disorder or myasthenia gravis.
3. Have a congenital disease such as acute coronary syndrome, cancer, or severe muscular or joint disease that affects the ability to walk continuously for at least 10 meters.
4. Be implanted with a pacemaker or electrical device.
5. Refuse or withdraw from the study.

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population included 164 people aged 50 - 59 years.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of sarcopenia | December2019
  participants with or without chronic lower back pain,

SECONDARY OUTCOMES:
The associated factors 1 | December2019
  age
The associated factors 2 | December2019
  body mass index
The associated factors 3 | December2019
  IPAQ
The associated factors 4 | December2019
  EQ-5D-5L
The associated factors 5 | December2019
  Congential diseases
The associated factors 6 | December2019
  Alcohol drinking
The associated factors 7 | December2019
  Cigarette smoking
The associated factors 8 | December2019
  Body muscular mass

CONTACTS AND LOCATIONS:
Overall Officials: Songsuda Roongsaiwatana, MD, Study Director — Ramathibodi Hospital
Locations (1):
- Physical medicine and rehabilitation, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu WT, Lee TM, Han DS, Chang KV. The Prevalence of Sarcopenia and Its Impact on Clinical Outcomes in Lumbar Degenerative Spine Disease-A Systematic Review and Meta-Analysis. J Clin Med. 2021 Feb 15;10(4):773. doi: 10.3390/jcm10040773. PMID 33671958